CLINICAL TRIAL: NCT00298740
Title: Reimplantation of Subjects With Implantable Insulin Pump Therapy
Brief Title: Medtronic MiniMed Implantable Insulin Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-05-01-08; RR00052
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Aventis U-400 Insulin (Experimental)
  Interventions: Device: Aventis U-400 Insulin

INTERVENTIONS:
Device: Aventis U-400 Insulin

SUMMARY:
This research is being done to find out whether subjects previously treated with the implantable insulin pump (IIP) therapy, and now taking insulin by injection, will benefit from re-implantation of IIP. The investigators will see if IIP causes more stable control of blood sugar, with fewer highs and lows. People with type 1 diabetes previously implanted with the MiniMed Implantable Pump (MIP) model 2000 at Johns Hopkins may join this study.

DETAILED DESCRIPTION:
If the participant joins the study and chooses to have a new pump implanted, the study is expected to last 12-15 months for each participant, and each participant will continue to be followed, with 3-monthly refills and research visits for as long as the pump lasts, until the participant chooses to withdraw, until the FDA approves the pump for regular care, or until the company stops supporting the pump. During the first 12-15 months of the study, there will be an estimated 13 clinic visits and one hospital stay for 2-3 days. The data collection visits will take about 30 minutes, and a continuous glucose monitor will be started. The participants will have a brief visit 3-4 days later to drop off the monitor. After this phase of the research, the participants will still be cared for with the implanted pump, having visits for refills and tests every 3 months. This long-term follow up will last until the participants choose to withdraw, the pump malfunctions, the FDA approves the pump for regular care, or the company no longer supports the pump. If the participants are no longer taking part in the study, the investigators will have the pump removed from their body.

ELIGIBILITY:
Inclusion Criteria:

* People with type 1 diabetes previously implanted with the MiniMed Implantable Pump model 2000 at Johns Hopkins may join this study.

Exclusion Criteria:

* Anyone not previously implanted with the MiniMed Implantable Pump model 2000 at Johns Hopkins.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-02 (Actual); Primary Completion 2009-09-24 (Actual); Study Completion 2009-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Saudek, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Witkowski CJ, Saudek C. The implantable peritoneal pump--a patient's perspective. J Diabetes Sci Technol. 2008 Jul;2(4):703-6. doi: 10.1177/193229680800200423. PMID 19885248
- [Background] Moore KB, Saudek CD, Greene A, Dackiw A. Implantable insulin pump therapy: an unusual presentation of a catheter-related complication. Diabetes Technol Ther. 2006 Jun;8(3):397-401. doi: 10.1089/dia.2006.8.397. PMID 16800761

RESULTS

PARTICIPANT FLOW:
Groups:
- Aventis U-400 Insulin: Aventis U-400 Insulin
Period: Overall Study
Arm/Group | Aventis U-400 Insulin
Started | 12
Completed | 3
Not Completed | 9
Not completed — Lack of Efficacy | 6
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Aventis U-400 Insulin
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Glucose Control as Assessed by Mean Glucose Levels
Time Frame: End of study, approximately 5 years
Population: It is unclear whether data was collected. No data is available and exhaustive searching has yielded no person with historical knowledge of this study or access to any data. Information obtained in other sections was from Regulatory records retrieved from long-term storage. This study closed in 2009 and the Principal Investigator is deceased.
Arm/Group | Aventis U-400 Insulin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Aventis U-400 Insulin
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aventis U-400 Insulin (N=12)
Death (Cardiac disorders) | 1 (1) — Heart Attack
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aventis U-400 Insulin (N=12)
Rectal hemorrage (Gastrointestinal disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 3 (3)
Hypoglycemia (Endocrine disorders) | 2 (2)
Left lower quadrant pain (Gastrointestinal disorders) | 1 (1)
Right groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Poison ivy (Skin and subcutaneous tissue disorders) | 1 (1)
Cataract surgery (Surgical and medical procedures) | 1 (1)
Pump stopped (Product Issues) | 1 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gall bladder surgery (Surgical and medical procedures) | 1 (1)
Adhesive capsulitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Swollen abdomen (Gastrointestinal disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lyme disease (Infections and infestations) | 1 (1)
Pump explant (Product Issues) | 6 (6)
High insulin antibodies (Immune system disorders) | 1 (1)
Diabetic ketoacidosis (Endocrine disorders) | 1 (1)
External Otitis (Eye disorders) | 1 (1)
Changed site location (Product Issues) | 1 (1)
Right ankle surgery (Surgical and medical procedures) | 1 (1)
Hyperglycemia (Endocrine disorders) | 3 (3)
Pump site infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes